CLINICAL TRIAL: NCT00817570
Title: Evaluation of Balance Reactions of Transfemoral Amputees Using the Virtual
Brief Title: Evaluation of Balance Reactions of Transfemoral Amputees Using the Virtual Analysis System
Status: Suspended | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Siev- Ner Itzhak, Sheba Medical Center
Other Study IDs: SHEBA-5610-08-IS-CTIL
Record Dates: First submitted 2009-01-04; First posted 2009-01-06 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Balance
Keywords: Trans Femoral Amputees Balance Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Transfemoral Amputees using the C- Leg knee.
- 2: Transfemoral Amputees using a Multiaxial Knee.
- 3: Able bodied.

SUMMARY:
The purpose of this study is to test and compare the balance reactions of Tranfemoral Amputees and able bodied subjects in response to perturbations given by a highly advanced Virtual Reality system.

ELIGIBILITY:
Inclusion Criteria:

* Transfemoral Amputees, walking without any assistive device, at least one year.

Exclusion Criteria:

* Amputees who suffer from a Neurological Injury/ disease that has implication on balance control.
* Amputees who suffer from Orthopedic Injury that has implication on balance control.
* Amputees who suffer from Cardiology disease that has implication on balance reactions.

Ages: 20 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Transfemoral Amputees and Able bodied.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel